CLINICAL TRIAL: NCT06296693
Title: Diagnostic Accuracy of Pocket-size Lung Ultrasound for Etiological Definition of Pneumonia and Surveillance of Complications in Children Hospitalized: a Prospective Diagnostic Cohort Study
Brief Title: Diagnostic Accuracy of Pocket-size Lung Ultrasound in Pneumonia Etiology and Complications in Hospitalized Children
Acronym: POCUS-L
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Universitário de Santo António (Other)
Responsible Party: Principal Investigator, Sara Monteiro, Dr., Centro Hospitalar Universitário de Santo António
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023.062(051-DEFI/053-CE)
Record Dates: First submitted 2023-12-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pneumonia; Pneumonia, Viral; Pneumonia, Bacterial
Keywords: bacterial pneumonia; community-acquired pneumonia; chest radiograph; digital health; POCUS; viral pneumonia
MeSH Terms: conditions — Pneumonia; Pneumonia, Viral; Pneumonia, Bacterial; Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POCUS-L (Experimental): The investigators will study the diagnostic accuracy of a pocket-size POCUS device vs. CXR for the etiological diagnosis of CAP, in paediatric age. During 1 year, all children aged >12 months and <18 years admitted to the Paediatric Department with the diagnosis of CAP on admission will be included. At least 76 participants will be required. Two investigators will perform, independently, a POCUS at admission, daily during hospitalization, 15 days and 1 month after discharge. All children will also undergo a CXR upon admission and whenever necessary. A third investigator will classify the CXR independently. It will be used the General Electrics Vscan AirTM®, with Bluetooth connection to smartphone/tablet. It will be collected the systematized description of POCUS and CXR, sociodemographic, clinical and therapeutic variables.
  Interventions: Device: Pocket-size lung ultrasound for etiological definition of pneumonia and surveillance of complications in children hospitalized

INTERVENTIONS:
Device: Pocket-size lung ultrasound for etiological definition of pneumonia and surveillance of complications in children hospitalized — The investigators will study the diagnostic accuracy of a pocket-size POCUS device vs. CXR for the etiological diagnosis of CAP, in paediatric age. During 1 year, all children aged >12 months and <18 years admitted to the Paediatric Department with the diagnosis of CAP on admission will be included. At least 76 participants will be required. Two investigators will perform, independently, a POCUS at admission, daily during hospitalization, 15 days and 1 month after discharge. All children will also undergo a CXR upon admission and whenever necessary. A third investigator will classify the CXR independently. It will be used the General Electrics Vscan AirTM®, with Bluetooth connection to smartphone/tablet. It will be collected the systematized description of POCUS and CXR, sociodemographic, clinical and therapeutic variables.

SUMMARY:
1. Background and study aims Pneumonia is the leading infectious cause of death in children worldwide. Although the diagnosis is clinical, a chest radiograph (CXR) is often necessary to clarify it, exposing the patient to radiation. Ultrasound has been increasingly used in the evaluation of the lung parenchyma without exposing patients to radiation. The pocket-size Point-of-Care Ultrasound (POCUS) can be used at the patient's bedside proving comfort and saving time. Evidence suggests that ultrasound can detect CAP (community-acquired pneumonia) in children with similar accuracy and reliability as CXR. However, few studies evaluated the ability to distinguish the aetiology of pneumonia and none used a pocket-size POCUS device. This study aims to assess, for the first time, the diagnostic accuracy of a pocket-size POCUS device for the etiological diagnosis of CAP vs. CXR, in paediatric ages. Secondarily, the investigators intend to evaluate the correlation between CXR image vs. ultrasound, the correlation between clinical progression and ultrasound images, and the diagnostic accuracy to detect complications.
2. Who can participate:

   The investigators will include, consecutively, all children aged >12 months and <18 years hospitalized to the Paediatric Department with the diagnosis of CAP on admission. The investigators will exclude children hospitalized with nosocomial pneumonia, with cystic fibrosis diagnosis or on long-term domiciliary ventilation.
3. What does the study involve:

   The diagnostic accuracy between POCUS and CXR in differentiating the type of pneumonia will be assessed. All participants will perform a POCUS at admission, daily during hospitalization, 15 days and 1 month after discharge. All children will also undergo a CXR upon admission and whenever necessary.
4. What are the possible benefits and risks of participating:

   Children will have a more frequent and serial assessment of CAP, which does not involve risks.
5. Where is the study run from:

   The study if from Centro Materno Infantil do Norte - Centro Hospitalar Universitário de Santo António, a tertiary paediatric referral centre.
6. When is the study starting and how long is it expected to run for:

The recruitment period is expected to start in January/2024 and end in January 2025.

DETAILED DESCRIPTION:
The investigators will perform a prospective diagnostic cohort study in a tertiary paediatric referral centre to study the diagnostic accuracy of a pocket-size Point-of-Care Ultrasound (POCUS) device vs. chest radiograph (CXR) for the etiological diagnosis of CAP, in paediatric age. During 1 year, all children aged >12 months and <18 years admitted to the Paediatric Department with the diagnosis of CAP on admission will be included. At least 76 participants will be required. Two investigators will perform, independently, a POCUS at admission, daily during hospitalization, 15 days and 1 month after discharge. All children will also undergo a CXR upon admission and whenever necessary. A third investigator will classify the CXR independently. It will be used the General Electrics Vscan AirTM®, with Bluetooth connection to smartphone/tablet. It will be collected the systematized description of POCUS and CXR, sociodemographic, clinical and therapeutic variables. Statistical analysis will be performed using SPSS® version 28.

This study won a competitive grant from MSD Portugal. The amount will be applied exclusively in the systematization and standardization of the POCUS technique with the guidance of an external consultant, in the statistical analysis, in the dissemination of results through participation in a national and international congress and in the creation of a task-force for the national implementation of this technique in paediatric services. The design, implementation, analysis, and dissemination of this stury will be independent from MSD Portugal and from the entire responsibility of the authors.

ELIGIBILITY:
Inclusion Criteria:

* Age >12 months and <18 years
* Hospitalization in the Paediatric Department
* CAP diagnosis on admission (based on the physician's clinical judgment, namely through clinical, analytical and/or CXR criteria)

Exclusion Criteria:

* Nosocomial pneumonia
* Cystic fibrosis diagnosis
* Long-term use of domiciliary ventilation.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
POCUS vs. CXR for the etiological diagnosis of CAP | From enrollment to the end of follow-up at 1 month
  Diagnostic accuracy of a pocket-size POCUS device for the etiological diagnosis of CAP vs. CXR, in paediatric ages.
  It will be classified as bacterial CAP in POCUS the association of lung consolidations, air bronchogram and shred sign. Viral CAP in POCUS will be considered in the presence of at least one: pleural abnormalities (irregularity or thickening), variable number (at least three) and coalescence of B-lines, multiple small subpleural consolidations.
  It will be classified as bacterial CAP in CXR when lung consolidations are present, represented as hypotransparencies areas that tends to occur initially in the peripheral subpleural lung and spreads centrally. Viral CAP in CXR will be considered in the presence of bilateral patchy hypotransparencies and diffuse areas of air space consolidation or interstitial lung disease.

SECONDARY OUTCOMES:
CXR image vs. ultrasound | From enrollment to the end of follow-up at 1 month
  Correlation between CXR image vs. ultrasound.
  The ultrasound findings will be compared with the radiological findings concerning at least one: lung consolidations, air bronchogram, pleural abnormalities, interstitial infiltrates.
Clinical progression and ultrasound images | From enrollment to the end of follow-up at 1 month
  Correlation between clinical progression and ultrasound images.
  Clinical progression will include three main symptoms: cough, shortness of breath and fever. POCUS findings over time (admission, daily during hospitalization, 15 days after discharge and 1 month after discharge) will include: lung consolidations, air bronchogram, shred sign, pleural abnormalities, variable number and coalescence of B-lines.
Complications | From enrollment to the end of follow-up at 1 month
  Diagnostic accuracy to detect complications.
  Complications will include the detection of at least one: pleural effusion, necrotizing pneumonia, lung abscess and pneumothorax on both POCUS and CXR.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Monteiro, Principal Investigator — Centro Hospitalar Universitário de Santo António

IPD SHARING:
Plan to Share IPD: No